CLINICAL TRIAL: NCT06924021
Title: Age-Related Macular Degeneration Benchmark Imaging Dataset (ABID)
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0059; Protocol Version 3/14/2025 (Other: UW Madison); A536070 (Other: UW Madison)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: screening; artificial intelligence; AI
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMD Benchmark Imaging Dataset Cohort: Study Procedures Include:
  * Patient history: demographics (age, sex, ethnicity, race), smoking history, family history of AMD
  * Physical exam: height and weight
  * Snellen best-corrected visual acuity (BCVA)
  * AMD classification (Beckman scale)
  Interventions: Other: Retinal Imaging

INTERVENTIONS:
Other: Retinal Imaging — Eligible participants will undergo one retinal imaging session of both eyes for the following:
  * Single field stereo color fundus photography (cFP) - pre and post dilation
  * Macular spectral domain-optical coherence tomography (SD-OCT)
  Other Names: Single field stereo color fundus photography; Macular spectral domain-optical coherence tomography

SUMMARY:
1000 participants from up to 25 international locations who are at least 50 years old with either healthy eyes or a diagnosis of Age-Related Macular Degeneration (AMD) will be consented to provide images of their eyes for a new dataset. This dataset is an important step in developing an Artificial Intelligence (AI) based screening tool for AMD.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a leading cause of blindness in the world. The early and intermediate stages of AMD progress to late stage resulting in vision loss due to either geographic atrophy or neovascular AMD. Preventive measures to reduce treatment burden and prevent blindness are important. While there are no approved therapies for early disease, active research is underway. However, advancing therapeutic trials for AMD prevention remains challenging due to the lack of primary care involvement in early-stage AMD diagnosis.

A clear need exists for a reliable screening tool, deployable in optometry or primary care facilities to identify those with an early stage of disease. While an Artificial Intelligence (AI) based screening tool would be an ideal solution, there are obstacles to its prospective validation due to difficulty in enrolling sufficient cases in a screening environment. A key step towards promoting this field lies in collecting a diverse dataset of multimodal imaging and providing a reference standard level 1 classification from a wide array of patients with AMD. Having such a benchmark dataset available for research purposes will empower the development and validation of AI models for AMD. This data can serve as the much-sought pathway to the rapid development of screening models, facilitating the referral of patients with the appropriate disease spectrum, and ultimately leading to the prevention of late AMD.

This is a prospective, cross-sectional, multi-center, observational study to collect and develop a meticulously curated and diverse AMD benchmark dataset, featuring reference standard level 1 classification and comprehensive annotation of images.

Study procedures include:

* Patient history: demographics (age, sex, ethnicity, race), smoking history, family history of AMD
* Physical exam: height and weight
* Snellen best-corrected visual acuity (BCVA)
* AMD classification (Beckman scale)

Eligible participants will undergo one retinal imaging session of both eyes for the following:

* Single field stereo color fundus photography (cFP) - pre and post dilation
* Macular spectral domain-optical coherence tomography (SD-OCT)

Due to the need for diversity in the dataset, sites need to represent a wide array of geographical locations. In addition, balancing will be done on enrolled participants with or without AMD including age, sex, and AMD level (worse eye selected as study eye).

ELIGIBILITY:
Inclusion Criteria:

* Participants greater than or equal to 50 years of age at time of signing Informed Consent Form
* Willing to comply with all study procedures and sign the Informed Consent Form (ICF)
* Individuals with normal healthy eyes or diagnosed with any stage of Age-Related Macular Degeneration (treatment naïve patients with early, intermediate, or late AMD). The diagnosis and eligibility review will be confirmed by Central Reading Center.

Exclusion Criteria:

* Therapeutic treatment for any type of AMD, in either eye. Supplements, such as AREDS2 formula, are allowed.
* Unable to acquire adequate quality images, as evaluated by the Central Reading Center
* Severe vision loss requiring urgent surgery
* Contraindicated for acquiring retinal images due to narrow anterior chamber angles or hypersensitivity to light
* A systemic or ocular condition that in the opinion of the Investigator would preclude participation in the study
* Unwilling to sign informed consent form
* Currently or previously enrolled in an interventional AMD clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 1000 participants from up to 25 sites in the United States, Europe, Asia, South America, Africa, and Australia will be enrolled and balanced by age, sex, and AMD level (worse eye selected as study eye). Every region listed above may not be represented and additional regions/countries not listed above may be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
AMD Classification by Participant Count | up to 18 months
  A meticulously curated and diverse Benchmark dataset, featuring reference standard level 1 classification and annotated images for a wide range of AMD phenotypes is the primary outcome. Diversity of the dataset will in part be measured by classifying AMD status.
  The goal is to have:
  * 20% participants with no AMD
  * 30% participants with Early AMD
  * 30% participants with Intermediate AMD
  * 10% participants with Geographic Atrophy (GA)
  * 10% participants with Neovascular age-related macular degeneration (nAMD)
Geographic Location by Participant Count | up to 18 months
  A meticulously curated and diverse Benchmark dataset, featuring reference standard level 1 classification and annotated images for a wide range of AMD phenotypes is the primary outcome. Diversity of the dataset will in part be measured by geographic location. 1000 participants from up to 25 global sites will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Amitha Domalpally, MD, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (14):
- United States (7):
  - Bergstrom Eye Research LLC, Fargo, North Dakota
  - Erie Retina Research, Erie, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retina Consultants of Texas (Houston), The Woodlands, Texas
  - University of Utah - John A. Moran Eye Center, Salt Lake City, Utah
  - University Station Eye Care Clinic, Madison, Wisconsin
- Charles Research Center, Buenos Aires, Argentina
- Adelaide Eye and Retina Centre, Adelaide, Australia
- Centre Hospialier Intercommunal de Paradis (Centre Monticelli Paradis), Marseille, France
- University of Bonn - Department of Ophthalmology, Bonn, Germany
- India (2):
  - Sankara Nethralaya, Medical Research Foundation, Chennai, Tamil Nadu
  - Aravind Eye Hospital, Chennai, Tamil Nadu
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No